CLINICAL TRIAL: NCT07064954
Title: Auto-PLTS: The Effectiveness of Autologous, Cold-stored Platelets Collected 7-10 Days Before Cardiac Surgery for Avoidance of Allogeneic Transfusions: A Randomized Patient Preference Trial
Brief Title: Autologous Cold-stored Apheresis Platelets
Acronym: Auto-PLTS
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-5285
Record Dates: First submitted 2025-07-07; First posted 2025-07-15 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Bleeding; Platelets; Cardiopulmonary Bypass; Cardiac Surgery
Keywords: Autologous Blood Donation
MeSH Terms: conditions — Hemorrhage | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Auto-PLTS is a single-centre trial that uses a randomized, patient preference design. Patients who agree to participate in the randomization stream will be assigned to the two study arms by random allocation. Those who do not consent to randomization but agree to participate in the patient preference stream will be assigned to their preferred arm of the study.
Who Masked: Outcomes Assessor
Masking Description: All safety outcomes will be collected by blinded research staff and reviewed by blinded assessors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Patients in the intervention group will undergo autologous collection of 2 units of apheresis platelets 7-10 days before surgery during their preadmission visit. The collected autologous platelets will be cold-stored at 1-6°C until the time of surgery. Patients will receive their own autologous platelets during or after surgery in response to excessive bleeding in the setting of low platelet count or function.
  Interventions: Biological: Autologous Cold-Stored Platelets
- Control Group (Active Comparator): Patients in the control group will receive standard, Health Canada approved, allogeneic platelets supplied by the Canadian Blood Services (stored at room temperature for up to 7 days) during or after surgery in response to excessive bleeding in the setting of low platelet count or function.
  Interventions: Biological: Allogeneic Room Temperature-Stored Platelets (Standard of Care)

INTERVENTIONS:
Biological: Autologous Cold-Stored Platelets — Two units of autologous platelets will be collected via an apheresis machine that draws blood from an intravenous (IV) line over 1-2 hours, isolates and leukoreduces the platelets by centrifugation and returns the remaining blood back to the patients. Collected autologous platelets will be stored at 1-6℃ without agitation until they are needed during or after surgery or 14 days have elapsed since their collection, after which they will be destroyed as per standard institutional procedures for expired blood products. For the first two platelet orders within 24 hours of cardiopulmonary bypass (CPB) termination, patients will receive their autologous cold-stored platelets. For the third and subsequent doses, patients in the intervention group will receive allogeneic room temperature-stored platelets (standard of care).
  Arms: Intervention Group
Biological: Allogeneic Room Temperature-Stored Platelets (Standard of Care) — Allogeneic platelets will be collected by Canadian Blood Services as per their standard operating procedures. Room temperature stored platelets will be stored at 20-24°C with constant agitation for up to 7 days as per current practices. For any platelet orders within 24 hours of cardiopulmonary bypass (CPB) termination, patients in the control group will receive allogeneic platelets as per usual care.
  Arms: Control Group

SUMMARY:
The Auto-PLTS Study is a single-centre trial performed at Toronto General Hospital (TGH) that uses a randomized, patient preference design. The recent introduction of cold-stored platelets with a shelf-life of 14 days into clinical practice has made it possible to offer autologous apheresis platelet predonation to patients undergoing elective cardiac (and other high-blood-loss) surgeries while allowing sufficient time to recover platelet count before surgery. The Auto-PLTS Study is designed to assess whether replacing allogeneic platelets with autologous platelets will improve patient outcomes and benefit the healthcare system by reducing the burden on allogeneic platelet supply. The study is also designed to determine whether patients are willing to donate autologous platelets 7-10 days prior to surgery.

ELIGIBILITY:
Inclusion Criteria:

Adult (≥18 years old) patients who meet all following criteria:

1. Undergoing elective complex cardiac surgery consisting of at least one of the following:

* Repair or replacement of more than one valve (i.e., multiple valves)
* Repair or replacement of any segment of aortic arch
* At least two of any combination of coronary artery bypass grafting (CABG), valve repair/replacement, or aorta (ascending/arch) repair/replacement
* Complex adult congenital repair

Exclusion Criteria:

Patients who meet any of the following criteria are not eligible for the study:

1. Seven days or less from recruitment to surgery (as there will not be sufficient time from platelet donation to surgery for patients to recover their platelet count)
2. Patient factors that preclude platelet donation or increase risk of adverse events after donation, including any of the following:

   * Poor intravenous access
   * Low baseline platelet count (≤150,000 x106/L)
   * Low baseline hemoglobin (<100 g/L) (since approximately 50 mL of red blood cells are lost with each unit of apheresis platelet collection)
   * Inability to tolerate fluid shifts during donation (i.e., severe aortic stenosis with valve area <0.7 cm2, or left main coronary artery stenosis >80%, or left ventricular ejection fraction <30%)
   * Increased risk of bacterial contamination of collected units (i.e., active infection, on antibiotics, dental procedure <72 hours before donation)
   * Attending clinicians deem the patient ineligible for autologous predonation
   * Known positivity for active infectious blood-borne disease (HIV, HCV, HBV, HTLV, Syphilis)
3. Highly specialized procedures such as insertion or removal of ventricular assist devices or repair of thoracoabdominal aneurysm
4. Any history of congenital or acquired bleeding disorder (including any type of thrombocytopenia or platelet refractoriness due to anti-platelet and anti-HLA antibodies or requirement for specially matched platelets)
5. On any anticoagulant or antiplatelet medications, excluding ASA, that cannot be stopped at least 7 days before donation (72 hours for NSAIDs)
6. Refusal of allogeneic blood products due to religious or other reasons
7. Known or suspected pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint | up to 24 hours after termination of cardiopulmonary bypass (CPB)
  The incidence of allogeneic platelet transfusion during the treatment period

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto General Hospital - University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No